CLINICAL TRIAL: NCT02607878
Title: Automated Pupillometry for Coma Prognostication After Cardiac Arrest
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: Erasme University Hospital (Other); Azienda Ospedaliera San Gerardo di Monza (Other); Lund University Hospital (Other); University Hospital, Grenoble (Other); Catholic University of the Sacred Heart (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Cochin University Hospital, Paris (Unknown); Charite University, Berlin, Germany (Other); Centre Hospitalier du Luxembourg (Other)
Responsible Party: Principal Investigator, Mauro ODDO, Médecin adjoint, PD-MER I, Centre Hospitalier Universitaire Vaudois
Other Study IDs: 432/14
Record Dates: First submitted 2015-11-02; First posted 2015-11-18 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Cardiac Arrest; Comatose
Keywords: Cardiac arrest; Coma; Prognosis; Automated pupillometry; EEG; Evoked potentials; Targeted Temperature Management (TTM)
MeSH Terms: conditions — Heart Arrest; Coma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Background: Sedation and therapeutic hypothermia (TH) delay neurological responses and might reduce the accuracy of clinical examination to predict outcome after cardiac arrest (CA). Electroencephalography (EEG) and somato-sensory evoked potentials (SSEP) might significantly improve prognostication of post-CA coma, however, EEG and SSEP are not always available and require specific expertise for their interpretation. Automated video pupillometry is a novel electronic device that contains an infrared light camera which enables to measure quantitatively the percentage of pupillary reaction to a calibrated light stimulation. In a recent study of a cohort of comatose CA survivors (n=50 patients) it was found that quantitative PLR was more accurate than standard PLR (manual pen light) in predicting 3-month outcome, irrespective of temperature and sedation, and had comparable prognostic accuracy than electrophysiological exams, including electroencephalography (EEG) and somato-sensory evoked potentials (SSEP).

Aim of the study: In light of these promising results, the investigators would like to confirm the prognostic value of quantitative PLR in a large multicenter cohort of comatose post-CA patients.

Design of the study: Prospective, multicenter, observational outcome trial.

DETAILED DESCRIPTION:
Study: Prospective, multicenter study. The study will be double-blinded, i.e. the clinician/nurse performing the tests will not be involved in patient care and clinicians in charge of patients will not be aware of automated pupillometry data. Patient care will not be influenced by pupillometry.

Patient population:

The investigators plan to include 500 comatose post-CA patients. The centers have been selected based on their expertise and publication track record on the topic, and because they are actively involved in the Neurointensive Care section (NIC) of the European Society of Intensive Care Medicine (ESICM). The study will take place at the Department of Intensive Care of the participating centers.

Patients will be managed according to standards of post-resuscitation care and based on local algorithms for the treatment of post-CA coma.

Quantitative pupillary light reactivity (PLR, using the NeurOptics NPi-200 pupillometer) will be performed on ICU admission and then every 12 hours up to 72 hours after CA. At each time point, one measurement will be assessed on both eyes.

The primary variables for analysis will be the neurological pupil index (NPi) and the pupil size for both eyes. Standard PLR using a manual pen light will be performed simultaneously at each time point, as part of standard care.

EEG, SSEP and sampling for serum neuron specific enolase (NSE) will be performed at 24h and at 48-72h, according to local practices and as part of standard care.

The predictive value of NPi will be analyzed using the area under the receiving operator characteristics (ROC) curve, and compared to that of standard PLR, EEG, SSEP and NSE: sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), unweighted accuracy, with 95% binomial confidence intervals, will be calculated. Associations with outcome will adjusted for main baseline demographics (age, initial CA arrest rhythm, time from CA to tROSC), dose of sedation-analgesia and vaso-active agents, and the SOFA score, using a logistic regression model.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with coma after cardiac arrest (CA)
* Glasgow Coma Scale (at inclusion): ≤ 6
* Patients with CA due to ventricular fibrillation (VF) and non-VF (including asystole and pulseless electrical activity) rhythms
* Cardiac and non-cardiac causes of CA will be included

Exclusion Criteria:

* Age < 18 years
* Unable to obtain consent
* Follow-up unavailable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coma after cardiac arrest (CA)
Sampling Method: Probability Sample
Enrollment: 470 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Neurological outcome | 3-6 months
  Neurological outcome is assessed by a semi-structured telephone interview with the patient or the patient's relatives using the Glasgow-Pittsburgh Cerebral Performance Categories (CPC). The CPC result is then categorized as favorable outcome (CPC 1-2, including good recovery and moderate disability), vs. unfavorable outcome (CPC 3-5, including severe disability, vegetative state and death).

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Oddo, MD, Principal Investigator — CHUV, Lausanne University Hospital, Switzerland
Locations (10):
- Erasme University Hospital, Brussels, Belgium
- France (2):
  - University Hospital, Grenoble, Grenoble
  - Cochin Hospital, Paris
- Charite University, Berlin, Germany, Berlin, Germany
- Italy (2):
  - Azienda Ospedaliera San Gerardo di Monza, Monza
  - Catholic University of the Sacred Heart, Roma
- Centre Hospitalier du Luxembourg, Luxembourg, Luxembourg
- Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA), Amsterdam, Netherlands
- Lund University Hospital, Lund, Sweden
- CHUV, Lausanne University Hospital, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No